CLINICAL TRIAL: NCT07043101
Title: Feasibility and Effectiveness of Goal Driven Extended Reality for Lower Limb Rehabilitation: A Pilot Study
Brief Title: Feasibility and Effectiveness of Goal Driven Extended Reality for Lower Limb Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University at Albany (Other)
Collaborators: Sunnyview Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0312-3
Record Dates: First submitted 2025-05-09; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Gait Rehabilitation
Keywords: Inpatient Rehabilitation; Augmented Reality; Gait Rehabilitation; Lower Extremity Function; Extended Reality; Mixed Reality; Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vector Based Gait Rehabilation paired with Extended Reality (Experimental): Individuals receiving Vector-based therapy will also receive Extended Reality (XR) during Vector sessions. The Extended Reality consists of mobility based tasks spaced along the Vector track that are executed through the XR headset.
  Interventions: Other: Extended Reality based Gait Rehabilitation

INTERVENTIONS:
Other: Extended Reality based Gait Rehabilitation — XR headset augmenting traditional Vector based gait rehabilitation.

SUMMARY:
This pilot study will evaluate the feasibility and preliminary effectiveness of incorporating Extended Reality (XR) into the treatment of patients undergoing Lower Limb Rehabilitation (LLR) using the Vector Gait and Safety System. LLR requires repetitive motions over the span of weeks or months with the aim of restoring mobility. This duration of time poses challenges with motivation and increases the burden on the physical therapists. The use of XR in conjunction with conventional physical therapy could significantly increase motivation, along with providing therapists with new ways of tracking the patient's recovery. Pilot study results will be used to propose new and innovative approaches to physical recovery during inpatient rehabilitation, potentially increasing motivation, enhancing therapy participation, and reducing the overall time taken for recovery.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at Sunnyview Rehabilitation Hospital
* Receiving or scheduled to receive Vector-based gait training therapy
* At least 18 years of age at the time of enrollment Exclusion Criteria
* Unable to use the Vector due to contraindications for Vector use (>500 lb or <30 lb), external halo neck support, severe osteoporosis, uncontrolled diabetes, uncontrolled hypertension, unstable fractures)
* Unable to follow 2 step commands
* Vertigo or vision abnormalities contraindicated for MR use
* Unable to ambulate prior to current injury
* In the judgment of the clinician, is not a good fit for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Gait Speed | 2 months
  Establish the efficacy of integrating Extended Reality (XR) with Vector treatment sessions during inpatient rehabilitation by monitoring the change in gait speed over sessions.

SECONDARY OUTCOMES:
Patient Motivation | 2 months
  Track patient motivation over sessions as measured by post session survey response on a 5 point Likert Scale (1-Not motivated, 5 - Very motivated).
Patient Confidence | 2 months
  Patient confidence in their rehabilitation while using the XR system. Measured by collecting patient feedback on post session survey using a 5 point Likert Scale (1- Not confident, 5- Very confident)
Patient Satisfaction | 2 months
  Measure how satisfied patient is with their recovery using the XR system. Captured using post session survey question with a 5 point Likert Scale (1-Very dissatisfied, 5- Very satisfied).

OTHER OUTCOMES:
Ease of Use, Enjoyability and Comfort | 2 months
  How easy, enjoyable and comfortable the overall system was for patients to use. Captured through post session survey questions with a 5 point Likert Scale for each (1- Very difficult/Not enjoyable/ Very uncomfortable, 5 - Very Easy/Very Enjoyable/Very comfortable).
End of study patient feedback | 2 months
  Feedback regarding challenges/difficulties, enjoyability, frustrations, and general suggestions. Collected post rehabilitation via a questionnaire.
Patient perceived effectiveness and challenge level | 2 months
  Effectiveness of XR session for patient rehabilitation, along with challenge posed via each task for the patient. Collected via post session survey questions with a 5 point Likert Scale (1-Not Effective/Much more challenging, 5- Very effective/Not challenging at all)

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnyview Rehabilitation Hospital, Schenectady, New York, United States

IPD SHARING:
Plan to Share IPD: No